CLINICAL TRIAL: NCT00613431
Title: A Randomized, Placebo-Controlled, Single Ascending Dose Study To Assess The Safety, Tolerability and Pharmacokinetics Of CS-8080 In Healthy Volunteers
Brief Title: Effects of CS-8080 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Karen Brown Ph.D. Associate Director, Experimental Medicine, Daiichi Sankyo Pharma Development
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS8080-A-U101; CS8080-A-U101
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2008-12

CONDITIONS: Healthy
Keywords: pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 6 dose groups, 9 subjects on active, 3 subjects on placebo in each group
  Interventions: Drug: CS8080
- 2 (Placebo Comparator): 3 subjects on placebo in each group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CS8080 — CS-8080 tablets will be administered once daily at doses of 1, 3, 10, 20, 50 and 100 mg.
  Arms: 1
Drug: Placebo — Some subjects will receive matching placebo instead of CS-8080.
  Arms: 2

SUMMARY:
The main purposes of this study are to assess the safety and measure the pharmacokinetics of CS-8080 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria Healthy men and/or women, aged 18 to 45 years inclusive.

* Women must be of non-child bearing potential, ie, either:Surgically sterile (ie, bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing), or Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing, with an FSH level at screening of > 40 mIU/mL.
* All women must have a negative serum pregnancy test at screening and within 48 hours before dosing.
* Body Mass Index (BMI) of 19 to 30 kg/m2 inclusive.
* Good health as determined by the absence of clinically significant deviation from normal, based on medical history, physical examination, laboratory reports, and 12 lead ECG, as deemed by the Investigator, prior to enrollment.
* Able to understand and willing to comply with all study requirements, and willing to follow the study medication regimen.
* Willing and able to give a written informed consent.
* Negative urine test for drugs of abuse and alcohol at screening and check-in.
* Negative result for HIV antibody, hepatitis B surface antigen, and hepatitis C antibody at screening.

Exclusion Criteria

* Any history of drug abuse.
* History of alcohol addiction during the 2 years prior to Day 1.
* History of significant allergic response to any drug except penicillin.
* History or current evidence, as determined by the Investigator, of psychiatric or emotional problems which would invalidate giving informed consent or limit the ability of the subject to comply with study requirements.
* History or current evidence of clinically significant cardiac, hepatic, renal, pulmonary, endocrine, neurologic, infectious, gastrointestinal (ie, any condition which may affect drug absorption), hematologic, or oncologic disease as determined by the Investigator after reviewing screening history, physical examination, laboratory test results, and 12-lead ECG.
* History or current alcoholic or non-alcoholic liver disease or liver steatosis.
* History of prostate disease or prostatitis.
* Subjects with a history of congenital Long QT Syndrome (LQTS), a history of surviving a near-drowning episode, or a history of any form of syncope or loss of consciousness.
* Subjects with QTc interval duration >450 msec obtained as an average from the ECG machine readings on the triplicate ECG (3 readings in rapid succession and not more than 2 minutes apart) taken at screening, after at least 10 minutes of quiet rest in a supine position.
* Subjects with abnormal ECG waveform morphology on any of the ECGs from the screening triplicate that would preclude accurate manual measurement of the QT interval duration.
* Need for any concomitant medication.
* Prestudy medication use as specified in Section 6.2.1.
* Consumption of any food or beverages containing grapefruit from 7 days prior to Day 1 through study completion.
* Consumption of foods or beverages containing alcohol from 24 hours before check-in through discharge from the clinic.
* Blood donation or significant blood loss within the 56 days before Day -1.
* Plasma donation within 7 days before Day -1.
* Participation in another investigational new drug research study within the 30 days before Day 1.
* Use of tobacco products or nicotine-containing products (including smoking cessation aids, such as gums or patches) within the 6 months before Day 1.
* Relationship of the subject to the Investigator, any sub-investigator, pharmacist, study coordinator, or other staff directly involved in the conduct of the study, or employment by the Sponsor or contract research organization participating in the study.
* Screening laboratory values outside the range of normal values deemed clinically significant by the Investigator. Serum lipid tests, triglycerides, cholesterol (LDL, HDL and total cholesterol), liver function tests (ALT, AST, GGT, total bilirubin, LDH and ALP) and PSA must not exceed the upper limit of normal without permission of the Sponsor.
* Hemoglobin <12.0 g/dL at the screening visit.
* Shift work, defined as any work shifts, either regular or irregular, precluding sleep during the hours of 10 pm and 6 am, within 1 week prior to Day -2, and no more than 2 works shifts per week meeting the above criteria from 4 to 1 week prior to Day -2.
* Positive fecal occult blood test at screening.
* Familial relationship with any other study participant.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety assessed over the 5-day post-dose inpatient period and at a follow-up 1 week post-discharge. | 2 weeks
Single dose plasma pharmacokinetics of CS-8080 | 2 weeks

SECONDARY OUTCOMES:
Pharmacodynamic response to CS-8080, as assessed by mRNA levels to 24 h post-dose. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noveck, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Neptune City, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/